CLINICAL TRIAL: NCT01082887
Title: A Phase I/II Study of Immunotherapy With TIL (Tumor Infiltrating Lymphocytes) in Combination With Intra-tumoral Injections of Interferon Gamma-adenovirus (Ad-IFNg) in Patients With Stage IIIc or Stage IV Metastatic Melanoma (AJCC)
Brief Title: A Study of Immunotherapy With TIL (Tumor Infiltrating Lymphocytes) in Combination With Intra-tumoral Injections of Interferon Gamma-adenovirus (Ad-IFNg) in Patients With Stage IIIc or Stage IV Metastatic Melanoma (AJCC)(Protocol TIL-Ad-INFg)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/09/05-R; 2009-013087-38 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Melanoma
Keywords: Immunotherapy TIL (Tumor Infiltrating Lymphocytes); Intra-tumoral injection; Interferon gamma-adenovirus(Ad-IFNg); Metastatic melanoma; A stage IIIc/IV metastatic melanoma with nodal relapse; in transit metastasis; cutaneous unresectable metastases; visceral metastases
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TIL-Ad-INFg (Experimental)
  Interventions: Other: TIL-Ad-INFg

INTERVENTIONS:
Other: TIL-Ad-INFg — After verification of inclusion and non-inclusion criteria and after obtaining informed consent from the patients, a tumor sample will be taken for sterile production of TIL. Patients will receive intra-tumoral injections of Ad-INFg every 15 days from J-15 to M2, then every month from M3 to M11 or until disease progression. The Ad-INFg will be administered by intra-tumoral injection at a dose of 5x1010 vp (viral particles) per lesion. A maximum of 6 lesions will be treated simultaneously. They will also receive two infusion of TIL at M0 (Cycle 1) and M1 (Cycle 2) by intravenous infusion lasting 30 to 65 minutes followed by subcutaneous injections of IL2 from J1 to J5 and from J8 to J12 of each cycle.An evaluation of injected and not injected tumoral lesions including photographs will be realised at the pre-inclusion visit, J-15, M0 and every month until M12.

SUMMARY:
The main objective of this study is to evaluate the clinical and biologic toxicity of cell therapy by adoptive transfer of TIL in combination with intra-tumoral injections of Ad-INFg.

ELIGIBILITY:
Pre-Inclusion Criteria:

* Male or female patients ≥ 18 and ≤ 75 years of age
* Patients must have signed informed consent
* A negative pregnancy test for women with childbearing potential
* Patients with stage IIIc/IV metastatic melanoma (AJCC 6th edition) with nodal relapse, in transit metastasis, unresectable cutaneous metastases, visceral metastases except bone and brain metastases
* Presence of at least one lesion accessible for intra-tumoral injections of Ad-IFNg
* A negative brain scan, eliminating any brain metastases
* ECOG performance status of 0-2
* Adequate bone-marrow reserve, renal function and hepatic function as assessed by standard laboratory criteria
* Subjects affiliated to an appropriate social security system

Inclusion Criteria:

* Negative viral serology (HIV ½, p24 Ag, HTLV 1 / 2, B and C hepatitis)

Exclusion Criteria:

* For female : the patient is pregnant or lactating or not using contraception and proved by a negative pregnancy test
* Positive viral serology for HIV ½, p24 Ag, HTLV 1 / 2 or B and C hepatitis
* History or current manifestations of severe progressive heart disease (congestive heart failure, coronary artery disease, uncontrolled arterial hypertension, serious rhythm disorders or ECG signs of previous myocardial infarction)
* Any serious illness, acute or chronic, e.g. active infection requiring antibiotics, bleeding disorders or any other condition that requires concomitant medications not allowed during this study
* Presence of a second active cancer except in situ cervical cancer or skin carcinoma
* Intercurrent disease requiring a corticosteroid treatment or a treatment with interferon-α
* Any autoimmune disease including active diabetes mellitus or immunodeficiency. Vitiligo in not an exclusion criteria
* Uncontrolled thyroid dysfunction
* Concurrently participation in a biomedical research (drug or radiotherapy) within the month preceding inclusion
* Metastatic lymph node stage alone with an indication of lymphadenectomy
* Brain or bone metastases discovered by radiological examination during the inclusion assessment
* Surgically resectable metastases
* Ocular melanoma
* More than one line of chemotherapy for treatment of melanoma
* Chemotherapy, immunotherapy or radiotherapy within 4 weeks before baseline (6 weeks for nitroso-ureas and mitomycin C)
* Contraindication for the use of vasopressor agents
* Treatment with molecules in pre-marketing development or whose development is finished less than 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clinical and biological toxicity of combined treatment TIL, IL2 et Ad-INFg | 12 months
  The evaluation of clinical and biological toxicity of combined treatment including infusion of TIL associated with subcutaneous injections of low-doses of IL-2 and intra-tumoral injections of Ad-IFNg will be performed according to clinical and biological criteria defined by NCI (Common Toxicity Criteria - version 3.0, August 2006).

SECONDARY OUTCOMES:
Objective response rate | 12 months
  The evaluation of the objective response rate
Tumoral response | 12 months
  The evaluation of the tumoral response of injected lesions every month
Progression-free survival | 12 months
  The evaluation of the progression-free survival,
Overall survival | 12 months
  The evaluation of the overall survival
Immunological response | 12 months
  The evaluation of the immunological response

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte DRENO, Profesor, Principal Investigator — Nantes University Hospital; Gaëlle QUEREUX, Doctor, Study Chair — Nantes University Hospital; Anabelle BROCARD, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France